CLINICAL TRIAL: NCT05796947
Title: From Active to Palliative Care: Emotional Burden and Self Efficacy in Patients and Caregivers
Acronym: CACP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4776
Record Dates: First submitted 2023-02-17; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: End of Life
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate psychological dimensions in patients and caregivers in the transition phase from active to palliative care.

DETAILED DESCRIPTION:
After being informed about the study, all patient giving written informed consent will enrolled and evaluated at T0 through the General Self-Efficacy Scale (GSE), Resilience Scale (RS-14), Toronto Alexithymia Scale (TAS-20), Integrated Palliative Care Outcome Scale (IPOS) and Caregiver Inventory (CGI).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients who are not undergoing active treatments (OLT)
* Suitability of the patient for palliative care
* Ability to express informed consent

Exclusion Criteria:

* Age < 18 years
* Patient not eligible for palliative care (active treatments)
* Comorbidity factors that make enrollment impossible
* Inability to give informed consent
* Psychiatric disorders prior to the current pathology
* Severe speech impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers declared "OLT/Off Therapy" for whom a suitable/eligible evaluation request is made by the clinicians to the UOC of Palliative Care (enrolled after clinical and psychological evaluations by the multidisciplinary team).
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Psychological assessment of Alexithymia domain in patient and caregiver | Test administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Assessment of the emotional state of patient and caregiver at the time of transition from active care to palliative care. The evaluation will be done by Toronto Alexithymia Scale, TAS-20 (G.J. Taylor, R.M. Bagby, J.D.A. Parker, 1992) to measure patient's and caregiver's ability to explore and share emotions.
  TAS-20 is a self-assessment questionnaire on alexithymia. It provides a total score, and the score of three dimensions that define the construct of Alexithymia: difficulty in identifying feelings, difficulty in communicating feelings to others and externally oriented thinking (operative thinking).
  It consists of 20 items measured on a five-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). A total score ranging from 20 to 100 is measured, plus three scores relating to the three dimensions of alexithymia. Clinical cut-off is from 60 to 100.
Psychological assessment of caregiver's burden domain. | Test administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Assessment of the caregiver burden at the time of transition from active care to palliative care. Assessment will be done by the following instrument:
  - Caregiver Inventory, CGI-I (S. Serpentini et al., 2021) to measure the caregiver's burden.
  It is a self-report tool for assessing the caring burden, it measures the self-efficacy of the caregiver in different aspects of caregiving such as managing medical information, taking care of the patient, take care of ownself and manage difficult interactions/emotions.
  The scoring scale is a Likert-type scale with a ranging from 1 (not at all confident) to 9 points (totally confident). Range scoring is from 9 to 189. The higher the score, the higher will be the caregiver's emotional and care burden.
Assessment of patient and caregiver self-efficacy domain. | Test administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Analysis of the results of the General Self-Efficacy Scale (GSE). It is a 10-item self-report psychometric scale that aims to measure the level of perceived self-efficacy to face the difficulties that life presents. It is a 5-point Likert-type scale. Score range is between 10 and 50, higher scores mean higher levels of perceived self efficay.
Psychological assessment of patient's burden domain. | Test administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Assessment of the patient's burden at the time of transition from active care to palliative care. Assessment will be done by the following instrument:
  - Italian Integrated Palliative Outcome Scale (IPOS): widely used as a measure of patient-reported outcome. IPOS studies patients' primary concerns: common symptoms, patient and family distress, existential well-being, sharing feelings with family, information received, and practical concerns.
  IPOS includes 10 symptoms and 7 questions about emotional situations, spiritual concerns, and provision of information and support.
  Five answer options are possible for each question (score from 0 to 4; higher scores indicate greater burden).
  The overall IPOS score is the sum of the scores for each of the 17 questions. The overall IPOS score can therefore range from 0 to 68 (80 if the patient adds the three additional symptoms to the proposed list).

SECONDARY OUTCOMES:
Assessment of patient and caregiver resilience domain. | Test administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Analysis of the results of the Resilience Scale (RS-14). This scale has got 14 items. It is a 7-point Likert-type scale: from 1 (strongly disagree) to 7 (strongly agree) for each item. Higher scores mean higher levels of resilience tendency. Minimum score:14, maximum score: 98. Clinical Cut-Off: < 56 very low resilience; 57 to 64: low resilience; 65 to 73: adeguate resilience; 74 to 81: moderate resilience; 82 to 90: high resilience; < 91: very high resilience.
Psychological differences between patients with first diagnosis or disease recurrence in self efficacy (assessed by General Self-Efficacy Scale) and resilience (assessed by Resilience Scale) domains. | Test to patients are administred just once, at Time 0 (up to 5 days after the clinical decision about the suspension of active tratements, and subsequently activation of Palliative Care Unit consultation).
  Evaluation of any differences between the examined psychological domains for patients with a first diagnosis or with disease recurrence. Correlation between outcomes in the two groups (first diagnosis vs recurrence) will be done at the end of the study by statistical analisys between variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No